CLINICAL TRIAL: NCT01170949
Title: Randomised, Double-blind, Placebo-controlled Study
Brief Title: Efficacy and Safety of Miltefosine in Antihistamine Resistant Chronic Urticaria
Acronym: MIARCU
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study medication expired
Sponsor: Marcus Maurer (Other)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor-Investigator, Marcus Maurer, Professor Dr.Marcus Maurer, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MIARCU 01/2008; EudraCT Number: 2007-007657-31
Record Dates: First submitted 2010-01-12; First posted 2010-07-28 (Estimated); Results first posted 2016-12-26 (Estimated); Last update posted 2016-12-26 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Urticaria
Keywords: urticaria
MeSH Terms: conditions — Chronic Urticaria; Urticaria | interventions — miltefosine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Miltefosine (Experimental)
  Interventions: Drug: Miltefosine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Miltefosine — 50 or 100 or 150mg per day
  Arms: Miltefosine
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Randomised, double-blind, placebo-controlled study evaluating the effects of miltefosine on skin lesions in patients with treatment resistant chronic urticaria. Treatment resistance is defined by insufficient treatment response after a minimum of 1 week therapy with the maximum labelled dose of a non-sedating antihistamine. Eligible subjects will be enrolled at baseline 8 (+/- 1) days after screening. 75 Patients will be randomised in a 2:1 ratio to one of the following treatment groups as add-on to the ongoing therapy with a non-sedating antihistamine for treatment period of 4 weeks: 25 placebo and 50 active drug Efficacy and safety evaluations are done at baseline day 7, 14, 21 safety, only) and 28 (or end of treatment) and at day 56 (28 days after end of treatment).

ELIGIBILITY:
Inclusion criteria Informed consent signed and dated Outpatients with moderate to severe spontaneous CU defined by UAS of ≥15 (under the maximum labelled dose of a non-sedating antihistamine Resistant to standard treatment with antihistamines after a minimum of 7 days therapy with the maximum labelled dose of a non-sedating antihistamine (levocetirizine, cetirizine, fexofenadine, desloratadine, loratadine, ebastine, mizolastine Aged more than 18 years Reliable method of contraception for both women of childbearing potential as well as men during the study and 3 months thereafter. A highly effective method of birth control is defined as those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, some IUDs, sexual abstinence or vasectomised partner.

Exclusion Criteria:

Pregnancy or lactation Participation in another clinical trial within the last 30 days Body weight ≤ 45 kg Subjects who are inmates of psychiatric wards, prisons, or other state institutions. Existing or planned placement in an institution after ruling according to § 40 passage 1 number 4 AMG (Arzneimittelgesetz).

Skin symptoms caused primarily by physical urticaria Urticaria vasculitis Known hypersensitivity to miltefosine Retinal pathology Leishmaniasis Gastrointestinal disturbances which may influence oral resorption (e.g. chronic diarrhoea diseases, congenital malformations or major surgical resection of gastrointestinal tract).

History within 5 years or presence of myocardial infarction or any other major cardiac disorder.

Serum-creatinine and/or BUN 1.5 times above the upper reference value GOT and/or GPT and/or alkaline phosphatase 3 times above the upper reference value).

Sjögren-Larsson-Syndrome. Malignancy within the last 5 years requiring chemotherapy or radiation therapy. Mental disorders that interfere with the evaluation of study end-points Drug or alcohol dependency Any other chronic or acute illness requiring systemic treatment which might have any influence on the outcome of the study in the 4 weeks before start of treatment and during the study (investigator's decision).

Immunodeficiency including HIV During the past 10 days before start of treatment and during the study Topical steroids H2 antihistamines Leukotriene antagonists H1 antihistamine other then basic therapy During the past 2 weeks before start of treatment and during the study Ketotifen Doxepin During the past 4 weeks before start of treatment and during the study Systemic corticosteroids UV therapy including PUVA Systemic immunosuppressives including corticosteroids, immunomodulators, immunostimulants During the past 12 weeks before start of treatment and during the study Astemizole Tranquilizers, antidepressants, sedatives, hypnotics, antiepileptics and other CNS active agents, except treatment with tricyclics that is stable for at least 12 weeks prior to screening and throughout the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2008-09; Primary Completion 2008-09 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Markus Magerl, MD, Principal Investigator — Charité University, Berlin
Locations (1):
- Charité University, Berlin, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Miltefosine; Placebo: Week 1 - 50 mg miltefosine or placebo Week 2 - 100 mg miltefosine or placebo (1 capsule in the morning and one in the evening),if evidence of intolerability dose had to be reduced to 50 mg, those patients received 50 mg until the end of the treatment period Week 3 - 150 mg miltefosine or placebo (3 capsules, one in the morning, one at lunch and one in the evening) if evidence of intolerability dose had to be reduced to 100 mg, those patients received 100 mg until the end of the treatment period
Period: Overall Study
Arm/Group | Miltefosine | Placebo
Started | 50 | 26
Completed | 43 | 22
Not Completed | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Miltefosine | Placebo | Total
Number analyzed (Participants) | 50 | 26 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 44 | 22 | 66
  >=65 years | 6 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.0 (12.4) | 42.6 (12.5) | 44 (24.9)
Gender [Count of Participants; unit: Participants]
  Female | 28 | 14 | 42
  Male | 22 | 12 | 34
Region of Enrollment [Number; unit: participants]
  Germany | 50 | 26 | 76

OUTCOME MEASURES:

1. Primary Outcome: Urticaria Activity Score (% Change From Baseline)
Description: The weekly UAS was calculated by adding the daily scores over one week. During the whole course of the study patients recorded the amount of wheals and the intensity of itching as well as the occurrence of swelling in ranges between 0 and 3. These daily scores were used to calculate urticaria activity scores (UAS) as follows: Daily UAS are calculated by adding the score points obtained for the symptom categories "number of wheals" and "intensity of pruritus". "Number of wheals" is scored as 0 = no wheals, 1 = some wheals (<20), 2 = moderate number of wheals (20-50), 3 = more than 50 wheals. "Intensity of pruritus" is scored as 0 = no itching; 1 = mild itching, not irritating; 2 = moderate itching, normal daily activity and sleep is possible; and 3 = severe itching, normal daily activity and sleep is impaired. The maximum score is 42.
Time Frame: Day 28
Population: ITT = 73
Measure: Mean (Standard Deviation); unit: percentage of UAS baseline
Arm/Group | Miltefosine | Placebo
Number analyzed (Participants) | 47 | 26
percentage of UAS baseline | -25.5 (38.2) | -10.1 (33.4)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at each Visit.
Arm/Group | Miltefosine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/26
Other Adverse Events (participants affected / at risk) | 44/50 | 17/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Miltefosine (N=50) | Placebo (N=26)
Abdominal discomfort (Gastrointestinal disorders) | 35 | 13
Nausea (Gastrointestinal disorders) | 14 (28) | 4
Vomiting (Gastrointestinal disorders) | 10 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No